CLINICAL TRIAL: NCT00736632
Title: Vitamin D, Insulin Resistance, and Cardiovascular Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); American Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201103002; R01HL094818 (NIH)
Record Dates: First submitted 2008-08-15; First posted 2008-08-18 (Estimated); Results first posted 2020-02-10 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-01

CONDITIONS: Vitamin D Deficiency; Insulin Resistance; Type 2 Diabetes Mellitus; Cardiovascular Disease; Hypertension
Keywords: Vitamin D; Insulin Resistance; Type 2 Diabetes Mellitus; Cardiovascular Disease
MeSH Terms: conditions — Vitamin D Deficiency; Insulin Resistance; Diabetes Mellitus, Type 2; Cardiovascular Diseases; Hypertension | interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Patients in the control group will receive placebo pills (instead of vitamin D) and calcium carbonate 500 mg twice daily.
  Interventions: Drug: Placebo
- Vitamin D (Active Comparator): Patients in the vitamin D group will receive cholecalciferol 4000 units daily and calcium carbonate 500 mg twice daily.
  Interventions: Drug: Vitamin D3

INTERVENTIONS:
Drug: Vitamin D3 — Cholecalciferol 4000 units orally daily Calcium carbonate 500 mg orally twice daily
  Other Names: Vitamin D
  Arms: Vitamin D
Drug: Placebo — Placebo pill orally daily Calcium carbonate 500 mg twice daily
  Arms: Placebo

SUMMARY:
In recent years, vitamin D has been shown not only to be important for bone and calcium metabolism but also for homeostasis of critical tissues involved in vascular disease in patients with diabetes. Epidemiological studies indicated the high prevalence of vitamin D deficiency among Type 2 DM patients and suggest an increased risk of cardiovascular disease and hypertension with low vitamin D levels. The objective of this proposal is to evaluate the effects of vitamin D replacement on blood pressure control and vascular disease in vitamin D deficient hypertensive patients with diabetes

DETAILED DESCRIPTION:
This is a double blinded, placebo controlled trial. Patients who meet the inclusion criteria will be randomized to placebo or 25(OH)D3, 4,000 IU/d orally for 16 weeks. Enrolled patients will be tested for 24h-blood pressure, brachial arterial blood flow, vascular inflammatory markers and macrophage inflammatory response to modified-lipoproteins at baseline, middle and at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* 25 (OH) vitamin D levels < 25 ng/ml
* Age 25 to 80 years
* Not on insulin for diabetes treatment
* HbA1c 5.5% -9.5%
* Mild/moderately increased blood pressure (systolic 120-160, diastolic 80-100) off BP medications

Exclusion Criteria:

* Pregnancy
* Patients with systolic >160 or diastolic >100 mmHg
* High urine calcium or history of recurrent kidney stones
* Cardiovascular disease
* Stage 3 or worse chronic kidney disease

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2006-05; Primary Completion 2019-01-13 (Actual); Study Completion 2019-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Bernal-MIzrachi, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington Universiy, St Louis, Missouri, United States

REFERENCES:
- See also: Washington University Endocrinology Department website — http://endo.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential participants will contact the principal investigator or research team through recruitment materials including emails to Washington University/Barnes Jewish/Children's staff, flyers, referrals through other physicians or the recruitment enhancement core, the Veterans Affairs Medical Center and Grace Hill Family Medical Center.
Pre-assignment Details: The third arm signed consent and are enrolled in the study but only for a single blood draw. They were not randomized and did not receive any intervention. No data was collected for any pre-specified primary or secondary outcomes from these participants.
Groups:
- Non-Intervention Blood Collection: Subjects without intervention will give a one-time blood sample for analysis of monocytes.
Period: Overall Study
Arm/Group | Placebo | Vitamin D | Non-Intervention Blood Collection
Started | 44 | 50 | 31
Completed | 44 | 50 | 31
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Non-intervention Blood Collection: Patients received no intervention. This is a one-time blood collection only.
- Total: Total of all reporting groups
Arm/Group | Placebo | Vitamin D | Non-intervention Blood Collection | Total
Number analyzed (Participants) | 44 | 50 | 31 | 125
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 41 | 44 | 24 | 109
  >=65 years | 3 | 6 | 7 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (8.8) | 56.1 (9.3) | 53.8 (13.2) | 54.3 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 28 | 24 | 69
  Male | 27 | 22 | 7 | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 28 | 23 | 25 | 76
  White | 15 | 27 | 5 | 47
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 44 | 50 | 31 | 125

OUTCOME MEASURES:

1. Primary Outcome: Hypertension (24h Blood Pressure, Central Blood Pressure, and Office BP)
Description: 24-hour blood pressure collected by ambulatory automated arm cuff, central mean arterial blood pressure (MAP) collected by non-invasive arterial tonometry and pulse wave analysis/pulse wave velocity, office blood pressure collected by manual aneroid sphygmomanometry.
Time Frame: 0, 2, and 4 months
Population: Occasional patients had missing blood pressure data or dropped out of the study prior to completion.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | Vitamin D
Number analyzed (Participants) | 44 | 50
mm Hg
  0 Month, Office SBP | 126.6 (14.3) | 131.1 (14.9)
  0 Month, Office DBP | 79.2 (10.7) | 78.9 (10.4)
  2 Month, Office SBP: number analyzed (Participants) | 43 | 50
  2 Month, Office SBP | 127.6 (16.4) | 133.2 (14.7)
  2 Month, Office DBP: number analyzed (Participants) | 43 | 50
  2 Month, Office DBP | 79.2 (10.5) | 79.9 (11.2)
  4 Month, Office SBP: number analyzed (Participants) | 44 | 48
  4 Month, Office SBP | 129.6 (16.9) | 132.7 (13.0)
  4 Month, Office DBP: number analyzed (Participants) | 44 | 48
  4 Month, Office DBP | 79.6 (9.5) | 77.9 (12.0)
  0 Month, Central MAP: number analyzed (Participants) | 41 | 48
  0 Month, Central MAP | 103.9 (9.3) | 107.2 (9.9)
  2 Month, Central MAP: number analyzed (Participants) | 42 | 48
  2 Month, Central MAP | 100.6 (9.0) | 107.8 (12.0)
  4 Month, Central MAP: number analyzed (Participants) | 42 | 47
  4 Month, Central MAP | 102.6 (9.3) | 105.2 (12.8)
  0 Month, Daytime MAP | 99.8 (6.3) | 101.6 (7.6)
  0 Month, Nighttime MAP: number analyzed (Participants) | 43 | 50
  0 Month, Nighttime MAP | 89.4 (8.2) | 92.2 (9.8)
  2 Month, Daytime MAP: number analyzed (Participants) | 38 | 45
  2 Month, Daytime MAP | 97.6 (10.7) | 101.7 (9.8)
  2 Month, Nighttime MAP: number analyzed (Participants) | 37 | 45
  2 Month, Nighttime MAP | 86.6 (9.7) | 94.0 (13.7)
  4 Month, Daytime MAP: number analyzed (Participants) | 44 | 46
  4 Month, Daytime MAP | 100.0 (10.7) | 99.1 (9.7)
  4 Month, Nighttime MAP: number analyzed (Participants) | 43 | 45
  4 Month, Nighttime MAP | 89.1 (12.0) | 90.3 (11.0)

2. Secondary Outcome: Brachial Artery Reactivity Testing
Description: Brachial artery response to hyperemia assessed by measuring brachial artery diameter every 30 seconds for 180 seconds after a 5-minute occlusion with arm cuff above systolic blood pressure, with response defined as maximal percentage increase above baseline.
Time Frame: 0, 2, and 4 months
Population: Some patients were unable to obtain adequate ultrasound images for BART analysis or did not show up for some visits
Measure: Mean (Standard Deviation); unit: percentage of dilation
Arm/Group | Placebo | Vitamin D
Number analyzed (Participants) | 44 | 50
percentage of dilation
  0 Month: number analyzed (Participants) | 44 | 43
  0 Month | 7.8 (5.9) | 8.6 (5.6)
  2 Month: number analyzed (Participants) | 42 | 44
  2 Month | 8.5 (6.6) | 7.5 (4.9)
  4 Month: number analyzed (Participants) | 44 | 38
  4 Month | 7.8 (4.6) | 7.8 (7.7)

3. Secondary Outcome: Macrophage Cholesterol Metabolism
Description: Macrophage uptake of labeled oxidized low density lipoprotein, assessed by the ratio of post-treatment cholesterol uptake to baseline uptake.
Time Frame: 0 and 4 months
Population: This analysis was only performed in a subset of patients.
Measure: Mean (Standard Deviation); unit: unitless (ratio)
Arm/Group | Placebo | Vitamin D
Number analyzed (Participants) | 15 | 11
unitless (ratio) | 1.01 (0.24) | 0.47 (0.072)

4. Secondary Outcome: Serum Calcium
Description: Serum calcium assessed by photometric assessment after calcium reaction with NM-BAPTA, then with EDTA
Time Frame: 0, 2, and 4 Month
Population: 1 placebo subject was unable to give samples at the 2 month visit, and 2 subjects were unable to give samples at the 4 month visit.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Vitamin D
Number analyzed (Participants) | 44 | 50
mg/dL
  0 Month, serum ca | 9.1 (0.5) | 9.1 (0.4)
  2 Month, serum ca: number analyzed (Participants) | 43 | 50
  2 Month, serum ca | 9.2 (0.4) | 9.1 (0.4)
  4 Month, serum ca: number analyzed (Participants) | 44 | 48
  4 Month, serum ca | 9.1 (0.4) | 9.3 (0.3)

5. Secondary Outcome: HbA1C
Description: HbA1c percentage assessed by turbidimetric inhibition immunoassay for hemolyzed whole blood
Time Frame: 0, 2, and 4 month
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Placebo | Vitamin D
Number analyzed (Participants) | 44 | 50
percentage
  HbA1c 0 month | 7.0 (1.2) | 7.0 (1.2)
  HbA1c 2 month: number analyzed (Participants) | 43 | 50
  HbA1c 2 month | 7.4 (1.8) | 6.9 (1.2)
  HbA1c 4 month: number analyzed (Participants) | 44 | 48
  HbA1c 4 month | 7.4 (1.9) | 7.0 (1.1)

6. Secondary Outcome: Vitamin D
Description: 25(OH) Vitamin D assess by liquid chromatography with tandem mass spectrometry
Time Frame: 0, 2, and 4 Month
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | Vitamin D
Number analyzed (Participants) | 44 | 50
pg/mL
  0 Month, Vitamin D | 46.1 (15.9) | 40.1 (11.9)
  2 Month, Vitamin D: number analyzed (Participants) | 43 | 50
  2 Month, Vitamin D | 37.7 (16.0) | 40.7 (11.3)
  4 Month, Vitamin D: number analyzed (Participants) | 44 | 48
  4 Month, Vitamin D | 44.5 (18.2) | 42.7 (17.1)

7. Secondary Outcome: hsCRP
Description: High sensitivity C-reactive protein assessed by particle-enhanced immunoturbidimetric assay
Time Frame: 0, 2, and 4 Month
Population: Several subjects were unable to give a sample at various time points.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Placebo | Vitamin D
Number analyzed (Participants) | 44 | 50
mg/L
  0 Month, hsCRP | 3.7 (3.0) | 6.0 (7.0)
  2 Month, hsCRP: number analyzed (Participants) | 43 | 50
  2 Month, hsCRP | 3.6 (2.9) | 5.9 (6.6)
  4 Month, hsCRP: number analyzed (Participants) | 44 | 48
  4 Month, hsCRP | 4.2 (4.0) | 6.7 (8.5)

8. Secondary Outcome: Fasting Glucose
Description: Serum fasting glucose assessed by hexokinase method
Time Frame: 0, 2, and 4 Month
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Vitamin D
Number analyzed (Participants) | 44 | 50
mg/dL
  0 Month, Fasting Glucose | 126.7 (34.5) | 123.3 (39.1)
  2 Month, Fasting Glucose: number analyzed (Participants) | 43 | 50
  2 Month, Fasting Glucose | 137.4 (57.6) | 124.9 (51.0)
  4 Month, Fasting Glucose: number analyzed (Participants) | 44 | 48
  4 Month, Fasting Glucose | 138.4 (55.2) | 128.7 (42.4)

9. Secondary Outcome: Urine Calcium to Creatinine Ratio.
Description: Urine calcium to creatinine ratio assessed by spectrophotometry
Time Frame: 0, 2 and 4 Months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/gm
Arm/Group | Placebo | Vitamin D
Number analyzed (Participants) | 44 | 50
mg/gm
  0 Month, ca to creatinine ratio | 69.8 (49.8) | 88.1 (94.8)
  2 Month, ca to creatinine ratio: number analyzed (Participants) | 43 | 50
  2 Month, ca to creatinine ratio | 102.3 (80.1) | 114.1 (62.5)
  4 Month, ca to creatinine ratio: number analyzed (Participants) | 44 | 48
  4 Month, ca to creatinine ratio | 89.9 (80.9) | 134.5 (106.5)

ADVERSE EVENTS:
Time Frame: The subjects in the placebo and vitamin D arm were monitored for adverse events from enrollment through completion which was over a course of 4 months.
Description: Adverse events were not collected or assessed from the the non-intervention blood collection arm.
Arm/Group | Placebo | Vitamin D
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/50
Other Adverse Events (participants affected / at risk) | 0/44 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-03): https://cdn.clinicaltrials.gov/large-docs/32/NCT00736632/Prot_SAP_000.pdf